CLINICAL TRIAL: NCT02081196
Title: Non-Invasive Reduction of Subcutaneous Fat Layer With an Alternative Treatment Parameter
Brief Title: CoolSculpting of the Flank With Alternate Treatment Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA13-005
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2020-09

CONDITIONS: Body Fat Disorder
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CoolSculpting of the Flank With Alternate Treatment Parameters (Experimental): Each subject served as their own control with 1 flank treated with CoolSculpting; the contralateral flank was untreated.
  Interventions: Device: The Zeltiq CoolSculpting System

INTERVENTIONS:
Device: The Zeltiq CoolSculpting System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of non-invasive subcutaneous fat layer reduction with an alternative treatment parameter.

DETAILED DESCRIPTION:
The study evaluated the use of the Zeltiq CooSculpting System for non-invasive fat removal in the flank.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects > 18 years of age and < 65 years of age.
2. Subject has clearly visible fat on the flanks, which in the investigator's opinion, may benefit from the treatment.
3. Subject has not had weight change exceeding 10 pounds in the preceding month.
4. Subject with body mass index (BMI) up to 30. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
5. Subject agrees to maintain his/her weight (i.e., within 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
6. Subject has read and signed a written informed consent form.

Exclusion Criteria

1. Subject has had a surgical procedure(s) in the area of intended treatment.
2. Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
3. Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 12 months.
4. Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
5. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
6. Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
7. Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
8. Subject is taking or has taken diet pills or supplements within the past month.
9. Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
10. Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
11. Subject is pregnant or intending to become pregnant during the study period (in the next 5 months).
12. Subject is lactating or has been lactating in the past 6 months.
13. Subject has a history of hernia in the areas to be treated.
14. Subject is unable or unwilling to comply with the study requirements.
15. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
16. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-02-18 (Actual); Primary Completion 2014-06-27 (Actual); Study Completion 2014-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Kilmer, MD, Principal Investigator — Laser and Skin Surgery Center of Northern California
Locations (3):
- United States (2):
  - Laser & Skin Surgery Center of Northern California, Sacramento, California
  - Dallas Plastic Surgery Institute, Dallas, Texas
- Arbutus Laser Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who seek reduction of fat in the flanks will be recruited from the general population.
Groups:
- CoolSculpting Intervention: CoolSculpting treatments were performed on one (1) flank in a single treatment visit. The contralateral flank served as the untreated control.
Period: Overall Study
Arm/Group | CoolSculpting Intervention
Started (Forty-five participants were enrolled. Subjects had 1 flank treated and 1 untreated.) | 45 (Treatment on one flank. Contralateral flank was untreated control.)
Untreated Control Flank (Each subject had one treated flank and one untreated flank.) | 45
Completed | 44 (One (1) subject was lost to FU.)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- CoolSculpting Intervention: CoolSculpting treatments were performed on one (1) flank in a single treatment visit.
Arm/Group | CoolSculpting Intervention
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 44.1 [23 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0
  Asian | 3
  Caucasian | 37
  Hispanic | 2
  Others | 3
Region of Enrollment [Number; unit: participants]
  Canada | 25
  United States | 20
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 24.1 [19.5 to 29.8]

OUTCOME MEASURES:

1. Primary Outcome: The Number of Device and/or Procedure-Related Adverse Events
Description: The number of device- or procedure-related adverse events will be tabulated. Adverse event reports are collected throughout the study from enrollment through the 16 week follow-up visit. The investigator determines if there is a relationship between the event and the study device or procedure.
Time Frame: Enrollment through 16 weeks post-treatment visit, which is approximately 5 months
Population: The safety population includes all subjects treated with CoolSculpting.
Measure: Number; unit: device or procedure-related AEs
Groups:
- CoolSculpting of the Flank With Alternate Treatment Parameters: Each subject served as their own control with 1 flank treated with CoolSculpting; the contralateral flank was untreated.
  Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration using the Zeltiq CoolSculpting System.
Arm/Group | CoolSculpting of the Flank With Alternate Treatment Parameters
Number analyzed (Participants) | 45
device or procedure-related AEs | 12

2. Primary Outcome: Change in the Fat Layer of the Treated Area as Measured by Ultrasound
Description: Change in the fat layer thickness will be calculated by comparison of pre-treatment and 16 week post-treatment ultrasound measurements taken in the area treated with the device, and in the untreated contralateral flank control area. The Sponsor's standardized techniques for obtaining ultrasound imaging will be used. Overall fat layer thickness changes were normalized for each subject by subtracting the change in control from the change in treated area to remove the influence of weight variations. Success is defined as, on average, at least a 1mm or greater reduction in fat layer thickness for the treated flank as compared to the untreated control flank. Results indicate the fat layer reduction in millimeters.
Time Frame: Pre-treatment and 16 weeks post-treatment
Population: Thirty-five subjects were included in the per-protocol analysis population: 1 subject was LTFU, 2 subjects did not complete the 16 week follow-up visit when ultrasonographer was present and 1 subject received an incomplete treatment. Six additional subjects had weight change greater than the protocol defined 5 pounds at the final follow-up visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CoolSculpting of the Flank With Alternate Treatment Parameters
Number analyzed (Participants) | 35
mm | -3.92 (2.45)
Statistical Analysis 1: Comparison: CoolSculpting of the Flank With Alternate Treatment Parameters; H0: μ(Control - Treated) < +1 versus H1: μ(Control - Treated) > +1; Test type: Other; Mean Difference (Net) = 4.13, 95% CI 2-sided [3.08 to 4.77], Standard Deviation 2.45 — Treatment Effect =Control Flank Change-Treated Flank Change such (a positive results indicates treated area had a larger reduction in fat thickness than control area, and a negative result indicates that a greater reduction was seen in control area)

3. Secondary Outcome: Proportion of Pre-treatment Images Correctly Identified.
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images. Images show both treated and untreated flanks. Reviewers will be practicing dermatologists or plastic surgeons. Reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Criteria for evaluable photos for the purposes of the independent review: subject completed treatments; subject has complete set of baseline photos and post-treatment photos; photos were taken using Zeltiq standard procedure. The expected success rate is 80% correct identification.
Time Frame: 16 weeks post-treatment
Population: The study population consisted of 45 participants. 1 subject was lost to follow-up; 1 subject had an incomplete treatment and photos of 1 subject were poor quality. Of the remaining 42 subjects, 7 did not maintain weight per protocol. 35 sets of subject photos were included in the analysis. Each image showed both treated and untreated flanks; both "arms" were included in the photo review.
Measure: Count of Units; unit: photos
Units Other Than Participants: photos
Arm/Group | CoolSculpting of the Flank With Alternate Treatment Parameters
Number analyzed (Participants) | 35
Number analyzed (photos) | 105
photos | 89
Statistical Analysis 1: Comparison: CoolSculpting of the Flank With Alternate Treatment Parameters; Test type: Other; sucess proportion = .8476, 95% CI 2-sided [.784 to .913]; Descriptive statistics (tabulation of Independent Panel Reviewer ratings) were used to analyze data

4. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction with the Zeltiq procedure as determined by the results of a subjects satisfaction questionnaire at the 16 week follow up visit. This questionnaire will be composed of 5-point Likert scale questions, as well as free-text responses.
Time Frame: 16 weeks post-treatment
Population: Of the 45 study participants, one subject received incomplete treatment and did not complete the questionnaire and one subject was lost to follow-up. Free text responses and inconclusive responses were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CoolSculpting of the Flank With Alternate Treatment Parameters
Number analyzed (Participants) | 43
Participants
  Procedure comfortable/very comfortable | 21
  Very visible to visible fat reduction | 37
  Positive overall effect | 34
  Somewhat to very different fit of clothing | 26
  Somewhat to very satisfied with procedure/results | 38
  Somewhat likely to likely to have another procedur | 39
  Very to somewhat likely to have same area treated | 24
  Would recommend procedure to a friend | 37

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through 131 days post-treatment.
Description: Protocol defined AE definitions: Adverse event is defined as any untoward medical occurrence in a subject, regardless of whether the event is related to the device. Adverse event data were aggregated for the study population as all subjects were treated with the Zeltiq System, with each subject having a treated flank and an untreated flank.
Groups:
- CoolSculpting of the Flank -Subjects With Systemic AEs: Each subject served as their own control with 1 flank treated with CoolSculpting; the contralateral flank was untreated.
- Flank Treated With CoolSculpting Group: One flank on each enrolled subject was treated with CoolSculpting.
- UnTreated Contralateral Flank: Each enrolled subject had one flank that was untreated, and no intervention was used.
Arm/Group | CoolSculpting of the Flank -Subjects With Systemic AEs | Flank Treated With CoolSculpting Group | UnTreated Contralateral Flank
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 7/45 | 12/45 | 0/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoolSculpting of the Flank -Subjects With Systemic AEs (N=45) | Flank Treated With CoolSculpting Group (N=45) | UnTreated Contralateral Flank (N=45)
Prolonged numbness in treatment area (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
First degree burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Post-treatment pain (General disorders) | 0 (0) | 3 (3) | 0 (0)
Cough and/or cold (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis and strep throat (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anxiety (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fractured heel (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No